CLINICAL TRIAL: NCT05545189
Title: Colorectal Polyp Histology Prediction by Artificial Ingelligence Method Based on NBI Colonoscopy Images.
Brief Title: Polyp Histology Prediction by Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Petz Aladar County Teaching Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PetzACTH2
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Polyp
Keywords: colorectal polyp,histology,artificial intelligence
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- colonoscopy group1: Polypectomy, histological examination, NICE classification and AIPHP analyzis will be performed 200 patients.
  Interventions: Diagnostic Test: colonoscopy,polypectomy
- colonoscopy group 2: Polypectomy, histological examination, NICE classification and AIPHP analyzis will be performed 200 patients
  Interventions: Diagnostic Test: colonoscopy,polypectomy
- colonoscopy group 3: Polypectomy, histological examination, NICE classification and AIPHP analyzis will be performed 200 patients
  Interventions: Diagnostic Test: colonoscopy,polypectomy
- colonoscopy group 4: Polypectomy, histological examination, NICE classification and AIPHP analyzis will be performed 200 patients
  Interventions: Diagnostic Test: colonoscopy,polypectomy
- colonoscopy group 5: Polypectomy, histological examination, NICE classification and AIPHP analyzis will be performed 200 patients
  Interventions: Diagnostic Test: colonoscopy,polypectomy
- colonoscopy group 6: Polypectomy, histological examination, NICE classification and AIPHP analyzis will be performed 200 patients
  Interventions: Diagnostic Test: colonoscopy,polypectomy

INTERVENTIONS:
Diagnostic Test: colonoscopy,polypectomy — polyp removal during colonoscopy

SUMMARY:
We have been developing artificial intelligence based polyp histology prediction (AIPHP) method to classify Narrow Band Imaging(NBI) colonoscopy images to predict the hyperplastic or neoplastic histology of polyps.

We plan to study colonoscopy polyp samples taken by polypectomy from 1200 patients.The documented NBI still images will be analyzed by the AIPHP method and by the NICE classification parallel.Our aim is to analyze the accuracy of AIPHP and NBI classification based histology predictions and also compare the results of the two methods.

DETAILED DESCRIPTION:
Background:

Colonoscopy with polypectomy or early colorectal neoplastic lesions (polyp) is a proven and widely accepted method of reducing colorectal cancer mortality rates.

Predicting histology prior to endoscopic colorectal polyp removal is useful especially for diminutive (1-5mm) and small (6-10mm ) polyps.

Evaluation of colorectal polyps using the narrow-band imaging (NBI) technique and the NBI International Colorectal Endoscopic (NICE) classification are useful to predict the histology during endoscopy.However, NBI and magnification based polyp histology prediction needs training and endoscopic experience. Morever , the final and objective diagnosis still requires histology.

Therefore,we have been developing arteficial intelligence-based polyp histology prediction (AIPHP) software to automatically evaluate the magnified NBI colonoscopy images aiming the histology prediction of polyps.

Materials and methods:

We plan to examine 1200 colorectal polyps obtained from patients. Polyps will be removed by traditional polypectomy or with mucosectomy.Endoscopic procedures and histological examinations performed at the participation hospitals. Colonoscopy will be performed with Olympus EXERA III CFHQ190I (Olympus ,Tokyo,Japan) high reolution NBI colonoscopes providing 65x optical magnification. Colorectal polyps will be detected first by high definition colonoscopy then by NBI at the optical maximum magnification (65x). All studied polyps will be photo-documented. The stored NBI photos were anelyzed by the NICE classification and AIPHP parallel system.

Histological examination methods:

We use WHO classification of colorectal polyps. The two -class classification will considere hyperplastic or neoplastic ((SSLs,tubular or villous adenomas, and invasive adenocarcinomas).

AIPHP software systtem:

The AIPHP software is based on the categorization of the vascular pattern and color of the polyps.The main steps of AIPHP software development will be the following: 1) feature vector calculation 2) training of classifier module, and 3) AIPHP classifier testing. Five features will be used by our AIPHP software.

ELIGIBILITY:
Inclusion Criteria:

* colorectal polyps removed by polypectomy

Exclusion Criteria:

* colorectal polyps with IBD

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colorectal polyps detected by colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-10-31 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Polyp histology accuracy by AI method | two weeks
  polyp histology prediction by AI

IPD SHARING:
Plan to Share IPD: No